CLINICAL TRIAL: NCT04356339
Title: US PROmyBETAapp2.0: Ascertaining Medication Usage and Patient-reported Outcomes (PROs) Via the myBETAapp™ in Patients With Multiple Sclerosis Treated With BETASERON® Using BETACONNECT™ Autoinjector
Brief Title: US PROmyBETAapp2.0: A Study to Learn More About the Medication Usage and Patient Reported Outcomes Via the myBETAapp in Medical Care of Patients With Multiple Sclerosis Treated With BETASERON Using BETACONNECT Autoinjector
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20756
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
Keywords: MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BETASERON: Participants with Multiple Sclerosis treated with BETASERON using BETACONNECT autoinjector and myBETAapp will be enrolled
  Interventions: Drug: Interferon-beta-1b (BETASERON, BAY 86-5046)

INTERVENTIONS:
Drug: Interferon-beta-1b (BETASERON, BAY 86-5046) — Using the BETACONNECT autoinjector and myBETAapp as prescribed by the physician

SUMMARY:
In this study researchers want to learn more about the medication usage behavior among multiple sclerosis (MS) patients treated with BETASERON using the myBETAapp. Multiple sclerosis (MS) is a disease in which the covering called "myelin" around the nerves of the central nervous system degenerate. MS is a lifelong disease therefore requiring continuous treatment to delay the disease progression and reduce the rate of relapse (the return of signs and symptoms of). BETASERON is an approved medicine used to reduce the relapse in patients with MS. It is injected into the tissue under the skin using BETACONNECT autoinjector, which automatically captures injection data including injection date, time, speed, and depth and uploads the data into paired myBETAapp. This allows patients to organize and track their progress and share the injection information with their physicians. The medication usage behavior to be collected in this study includes the elements to what extent

* taking medication matches the presciber's recommendation (adherence, compliance),
* treatment for the prescribed duration (persistence) is continued and
* injections were missed. Among MS patients treated with Betaferon using the myBETAapp the study will also collect information on the health-related quality of life , treatment satisfaction and satisfaction with treatment support.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Treated with BETASERON using the BETACONNECT autoinjector
* Registered with myBETAapp
* Provided electronic informed consent

Exclusion Criteria:

- There are no exclusion criteria for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: US patients aged ≥18 years diagnosed with Multiple Sclerosis (MS) and treated with BETASERON using the BETACONNECT autoinjector and registered with myBETAapp
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Compliance to therapy | Up to 6 months
  Compliance is defined as the the proportion of BETASERON administrations with the correct injection interval within some window. Windows will be set for each individual patient based on prescribed injection frequency.
Persistence of therapy | Up to 6 months
  Persistence to BETASERON using the BETACONNECT device will be measured as the number of days between the initial BETASERON administration and the earlier of the last BETASERON administration using the BETACONNECT device or before a minimum 60-day gap in therapy.
Adherence to therapy | Up to 6 months
  Adherence to BETASERON using the BETACONNECT device is a dichotomous variable (adherent or non-adherent) defined as receiving at least 80% of the expected number of injections during 6 months of treatment (or up to the point of early termination) as captured by the BETACONNECT device.

SECONDARY OUTCOMES:
Change in patient-reported health-related quality of life (HRQOL) | Up to 6 months
  Change in patient-reported health-related quality of life (HRQOL) will be collected via an online study-specific patient survey.
Patient satisfaction with the myBETAapp | Up to 6 months
  Patient satisfaction with the myBETAapp will be collected via an online study-specific patient survey.
Change in health status evaluated by EQ-5D-5L descriptive system | Up to 6 months
  EQ-5D-5L is a standardized measure of general health status. The EQ-5D-5L descriptive system consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), where respondents indicate their health state on each dimension based on 5 response options (no problems, slight problems, moderate problems, severe problems, and extreme problems).
Change in EQ-Visual Analog Score (EQ-VAS) | Up to 6 months
  The EQ-Visual Analog Score (EQ-VAS) allows respondents to rate their health on a 20 cm vertical, visual analog scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine' and provides a single quantitative measure of health.
Change in prescription and non-prescription medication usage | Up to 6 months
  Prescription and non-prescription medication usage will be collected via an online study-specific patient survey.
Number of relapses | Up to 6 months
Number of participants with treatment with corticosteroids due to relapses | Up to 6 months
Number of emergency room visits due to relapse | Up to 6 months
Number of hospitalizations due to relapse | Up to 6 months
Patient self-assessment | Up to 6 months
  Self-assessment includes assessment for mood, memory, vision, urinary symptoms. The assessment will be collected via an online study-specific patient survey.
Change in dose of BETASERON prescription | Up to 6 months
Change in frequency of BETASERON prescription | Up to 6 months
Patient satisfaction with the BETACONNECT autoinjector | Up to 6 months
  Patient satisfaction with the BETACONNECT autoinjector will be collected via an online study-specific patient survey.

CONTACTS AND LOCATIONS:
Locations (1):
- myBETAapp, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.